CLINICAL TRIAL: NCT05407766
Title: A Phase I Safety Study of Allogeneic Bone Marrow Derived MSCs for Refractory Perianal Fistulizing Crohn's Disease
Brief Title: Mesenchymal Stem Cells (MSCs) for Perianal Fistula
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: OSSM-001 will not be used in this clinical program.
Sponsor: Ossium Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OSSM-001-001-01
Record Dates: First submitted 2022-05-09; First posted 2022-06-07 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Rectal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 100M of OSSM-001 (Experimental): Single injection of mesenchymal stem cells at dose of 100M
  Interventions: Biological: OSSM-001
- 300M of OSSM-001 (Experimental): Single injection of mesenchymal stem cells at dose of 300M
  Interventions: Biological: OSSM-001
- Placebo (Placebo Comparator): Single injection of normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: OSSM-001 — Single injection of OSSM-001 at dose of 100M or 300M cells
  Arms: 100M of OSSM-001; 300M of OSSM-001
Other: Placebo — Single injection of placebo (saline)
  Arms: Placebo

SUMMARY:
OSSM-001 will be evaluated in a double blind, randomized phase I safety study of a single injection of 100 and 300 million bone marrow derived MSCs in 16 patients with refractory perianal fistulas in the setting of Crohn's disease. There will be 2 cohorts (100M and 300M MSCs); 8 subjects in each cohort; 6 subjects receiving the investigational product and 2 subjects receiving placebo (normal saline) in each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women 18-75 years of age with a diagnosis of unhealing perianal fistulas in the setting of Crohn's disease and must be on maximal standard of care therapy (e.g., antibiotics, 5-ASA, and immunomodulator, anti-TNF, anti-integrin, and anti-interleukin therapies) for at least six months duration.
* Presence of perianal fistula with maximum of two internal fistula tracts and a maximum of three external openings based on clinical assessment and MRI. Fistula must have been draining for at least 6 weeks prior to the screening visit.
* Medically refractory perianal fistulizing Crohn's disease (i.e., standard of care such as antibiotics, immunosuppressives)
* Have no contraindications to MR evaluations: e.g., pacemaker or magnetically active metal fragments, claustrophobia
* Ability to comply with protocol
* Competent and able to provide written informed consent
* Concurrent Crohn's-related therapies with stable doses corticosteroids, 5- ASA drugs, immunomodulators, anti-TNF therapy, anti-integrin and anti-interleukin therapies are permitted.
* A female participant and of childbearing potential must have a negative serum or urine pregnancy test at time of screening, and must not plan to become pregnant during the study.

Exclusion Criteria:

* Inability to give informed consent.
* Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
* Specific exclusions: Hepatitis B or C, HIV, Abnormal AST or ALT at screening
* History of cancer including melanoma (with the exception of localized skin cancers) in the past five years
* Received treatment with an investigational drug or device within 60 days of randomization or have not completed 5 half-life washout (whichever is later) for drugs or biologics. If the half-life of the product is not known, then subjects cannot be randomized within 6 months of investigation drug treatment.
* Participated in a cell therapy-based trial within 6 months before randomization
* Participated in Crohn's/ulcerative colitis or any fistulizing Crohn's study within 6 months before randomization
* Pregnant or breast feeding or trying to become pregnant.
* Presence of a rectovaginal or perineal body fistula
* Change in Crohn's immunosuppressive regimen prior to enrollment. Subjects should be on stable, maximal medical therapy for 4 months prior to enrollment.
* Uncontrolled intestinal Crohn's disease which will require escalation for medical therapy or surgery within 3 months of enrollment
* Severe anal canal disease that is stenotic and requires dilation or severe proctitis making difficult to the surgery
* A female or male participant unwilling to agree to use acceptable contraception methods during participation in study. Acceptable contraception methods include: Implants, injectables, combined oral contraceptives, an intrauterine device, a bilateral tubal ligation, a vasectomy, a vasectomized partner for female participant, double-barrier methods, and physical barrier if male participant is not vasectomized
* Associated perianal abscess(es).
* Laboratory exclusions: Serum creatinine levels >1.5 times the upper limit of normal (ULN). Total bilirubin >1.5 × ULN. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5.0 × ULN. Hemoglobin <10.0 g/dL for females or <11.0 g/dL for males. Platelets <75.0 × 109/L.
* Any contraindications to MRI or surgical or anesthetic procedure(s)
* Any major GI surgery or major perianal local surgery within 6 months of randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
OSSM-001 (100M dose) related adverse events as assessed by CTCAE v5.0 | 12 weeks
  To determine the safety of a single injection of 100M allogeneic bone marrow MSCs for the treatment of refractory perianal fistulizing Crohn's disease by assessing OSSM-001 related adverse events as assessed by CTCAE v5.0.
OSSM-001 (300M dose) related adverse events as assessed by CTCAE v5.0 | 12 weeks
  To determine the safety of a single injection of 300M allogeneic bone marrow MSCs for the treatment of refractory perianal fistulizing Crohn's disease by assessing OSSM-001 related adverse events as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Fistula healing assessed by radiographic (MRI) assessments for OSSM-001 (100M dose) | 12 weeks
  To assess fistula healing induced by the delivery of a single injection of 100M allogeneic bone marrow derived MSCs on refractory perianal fistulizing Crohn's disease using radiographic assessment (MRI) assessments.
  Complete healing defined as MRI with an absence of a fluid collection >2cm in 3 of 3 dimensions, lack of edema, inflammation, or sign of active inflammatory response. A remnant of scar of a fistula tract may remain.
  Partial healing defined as MRI with an absence of a fluid collection >2cm in 2 of 3 dimensions, lack of edema, inflammation, or sign of active inflammatory response. A remnant of scar of a fistula tract may remain.
  Lack of response defined as healing which does not meet the threshold for partial healing.
  Worsening disease defined as MRI with fluid collection >2cm in 2 of 3 dimensions, edema, inflammation, or sign of active inflammatory response. An increased number of tracts may be seen, or increased branching from the primary tract.
Fistula healing assessed by clinical assessments for OSSM-001 (100M dose) | 12 weeks
  To assess fistula healing induced by the delivery of a single injection of 100M allogeneic bone marrow derived MSCs on refractory perianal fistulizing Crohn's disease using clinical assessments.
  Complete healing defined as 100% cessation of drainage on clinical exam and with gentle finger compression.
  Partial healing defined as greater than or equal to 50% cessation of drainage on clinical exam with gentle finger compression.
  Lack of response defined as healing which does not meet the threshold for partial healing.
  Worsening disease defined as increased drainage on clinical exam.
Fistula healing assessed by radiographic (MRI) assessments for OSSM-001 (300M dose) | 12 weeks
  To assess fistula healing induced by the delivery of a single injection of 300M allogeneic bone marrow derived MSCs on refractory perianal fistulizing Crohn's disease using radiographic assessment (MRI) assessments.
  Complete healing defined as MRI with an absence of a fluid collection >2cm in 3 of 3 dimensions, lack of edema, inflammation, or sign of active inflammatory response. A remnant of scar of a fistula tract may remain.
  Partial healing defined as MRI with an absence of a fluid collection >2cm in 2 of 3 dimensions, lack of edema, inflammation, or sign of active inflammatory response. A remnant of scar of a fistula tract may remain.
  Lack of response defined as healing which does not meet the threshold for partial healing.
  Worsening disease defined as MRI with fluid collection >2cm in 2 of 3 dimensions, edema, inflammation, or sign of active inflammatory response. An increased number of tracts may be seen, or increased branching from the primary tract.
Fistula healing assessed by clinical assessments for OSSM-001 (300M dose) | 12 weeks
  To assess fistula healing induced by the delivery of a single injection of 300M allogeneic bone marrow derived MSCs on refractory perianal fistulizing Crohn's disease using clinical assessments.
  Complete healing defined as 100% cessation of drainage on clinical exam and with gentle finger compression.
  Partial healing defined as greater than or equal to 50% cessation of drainage on clinical exam with gentle finger compression.
  Lack of response defined as healing which does not meet the threshold for partial healing.
  Worsening disease defined as increased drainage on clinical exam.

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Munjal, MD, Study Director — Ossium Health, Inc.; Amy Lightner, MD, Principal Investigator — The Cleveland Clinic